CLINICAL TRIAL: NCT06874660
Title: Influence of Timing on Outcomes of Pancreaticoduodenectomy: Complications, Hospital Costs, and Length of Stay
Brief Title: Effects of Surgical Timing on Perioperative Clinical Outcomes in Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xinrui Zhu，MD, MD, The Third Affiliated Hospital of Soochow University
Other Study IDs: 2025-001
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pancreaticoduodenal; Fistula; Surgery Timing; Perioperative Complication
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: surgery before 12.00 pm
- 2: surgery before 12.00 pm

SUMMARY:
With the advancement of surgical techniques and the increase in pancreatic oncologic diseases, the volume of pancreaticoduodenal surgeries has been increasing year by year in our center, and multiple pancreaticoduodenal surgeries are often performed on the day of surgery. This study will compare the effect of pancreaticoduodenal surgery performed at different times on patient prognosis. This study plans to divide the patients into morning group, afternoon group, and night group through the start time of surgery, and this study plans to analyze subgroups such as laparoscopic pancreaticoduodenal surgery. The outcome indicators include perioperative complications such as pancreatic fistula, bleeding, abdominal infection, hospitalization cost, and length of hospital stay. The conclusions drawn from this study will suggest to surgeons whether pancreaticoduodenal surgery performed at different times of the day will have different outcomes for patients and will guide surgeons on the timing of pancreaticoduodenal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be required to sign an informed consent form;
2. Age 18-80 years, male and female;
3. ECOG Physical Status Score (PS Score) 0 or 1.
4. Pancreaticoduodenectomy at our center without contraindications related to the surgery.

Exclusion Criteria:

1. Pre-existing or concurrent other malignant tumors
2. Severe cardiopulmonary and renal dysfunction.
3. Autoimmune disease or history of immunodeficiency
4. Active infections and infectious diseases requiring systemic therapy.
5. History of psychotropic substance abuse, alcoholism or drug addiction.
6. Failure to meet the inclusion criteria as determined by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met the surgical guidelines for pancreaticoduodenectomy and underwent pancreaticoduodenectomy during the trial period
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
perioperative complication | perioperative
  pancreatic fistula; postoperative bleeding; abdominal infection; delayed gastric emptying

SECONDARY OUTCOMES:
Length of hospitalization | perioperative
  Length of admission to surgery; length of surgery; length of postoperative stay to discharge

OTHER OUTCOMES:
Cost of hospitalization | perioperative
  Cost of surgery; cost of postoperative medications; total cost of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Xinrui Zhu, Changzhou, Jiangsu, China